CLINICAL TRIAL: NCT02070393
Title: Breast-Sparing Proton Therapy for Hodgkin's Disease in Young Females Demonstrated By Positron Emission Tomograpy (PET) Scanning: A Pilot Study
Brief Title: Breast-Sparing Proton Therapy for Hodgkin's Disease
Acronym: Breast Sparing
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Closure of Indiana University Health Proton Center in December 2014
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IUHPTC-01
Record Dates: First submitted 2012-04-19; First posted 2014-02-25 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Hodgkins Disease
Keywords: Hodgkins Disease in Young Females; Breast Sparing Radiation Treatments
MeSH Terms: conditions — Hodgkin Disease | interventions — Protons

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Treatment using Protons (Experimental): 14 -24 Radiation Treatments (typically 1.5 - 1.8 cobalt-Gray equivalent per fraction for 14-24 treatments).
  Interventions: Radiation: Proton

INTERVENTIONS:
Radiation: Proton — 14-24 Radiation treatments using Protons
  Other Names: Breast sparing using proton beams

SUMMARY:
The purpose of this study is to drastically reduce unnecessary breast dose in young females with Hodgkin's Disease who require radiation therapy.

DETAILED DESCRIPTION:
According to the National Cancer Institute's Surveillance, Epidemiology, and End Results Program, there will be an estimated 8,490 new cases of Hodgkin's Lymphoma (HL) in the United States in 2010, with an estimated 1,320 deaths (Jemal, Siegel et al.). The unadjusted rates of 5 year overall survival are approximately 95%, and remain among the highest of all childhood and adult malignancies. With many children and young adults surviving into advanced age, the impetus has been to develop less toxic yet equally effective treatments. One of the main approaches taken over the last 25 years to minimize long-term treatment toxicity has been to limit the amount and volume of radiation received by patients. This pilot study continues along those lines, attempting to further refine the delivery of radiation therapy (RT) in order to avoid one of the most notorious long-term side-effects: secondary breast cancer.

Multiple studies investigating late toxicity in long-term survivors of pediatric Hodgkin's Lymphoma have shown the risk of breast cancer in young females receiving mediastinal radiation to be 50 times greater than their age-matched counterparts. The Late Effects Study Group, with a median follow-up of 17 years, reported a breast cancer incidence of 16% with a standardized incidence ratio of 55.5 (Bhatia, Yasui et al. 2003). Through utilization of breast-sparing proton therapy, we hope to provide young female patients with the benefits of radiation therapy while decreasing their risk of secondary breast cancer, thus increasing the therapeutic ratio.

In a prior computer-based, in-silico, dose planning study, utilizing the most basic beam orientation (a single PA beam), we showed that dose to breast tissue was reduced by a minimum of at least 80% with proton treatment compared to standard AP-PA photon treatment (in publication). Furthermore, dose to clinical target volume was maintained, and dose to other normal structures was statistically no worse. We now aim to validate these findings by verifying the beam range, in-vivo, via post-treatment combined Positron Emission Tomography-Computer Tomography (PET-CT) imaging in young females undergoing supra-diaphragmatic radiotherapy for Hodgkin's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age >/= 10 years old and < 30 years old
* Pathologically confirmed classical Hodgkin's Lymphoma
* At least one site of disease located above the diaphragm
* Signed study-specific consent prior to initiation of therapy
* Women of child-bearing potential must have a negative pregnancy blood test within 7 days of starting protocol therapy.

Exclusion Criteria:

* Previous radiation therapy to any part of the body.
* Parenchymal lung involvement at initial presentation or any patient that may need whole lung irradiation as per institutional guidelines.
* Lymphocyte predominant histology not eligible.
* Significant infection or other coexistent medical condition that would preclude protocol therapy such as:

  * History of HIV/AIDS
  * History of collagen Vascular Disease
  * Symptomatic congestive heart failure
  * Unstable angina pectoris or myocardial infarction within 6 months
  * Uncontrolled hypertension (systolic blood pressure > 160 mm Hg or diastolic blood pressure > 100 mm Hg on 2 consecutive measurements separated by 1 week).
  * History of uncontrolled diabetes
  * Psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements

Ages: 10 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Comparative DVH data for delivered proton plan and accompanying photon plan for target volume and normal tissues. | 12 months
  Dose-volume histogram data from both the delivered proton plan and the accompanying photon plan for target volumes and normal tissues, including:
  • Breast, heart, lung, thyroid, parotid glands , esophagus, spinal cord, *liver, *kidneys,

SECONDARY OUTCOMES:
Treatment toxicity and disease control of proton therapy for the treatment of pediatric Hodgkin's Lymphoma. | 3 - 60 Months
  1. Acute toxicity as per CTCAE v4.0
  2. Local, regional, and distal control of the disease at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Buchsbuam, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Health Proton Therapy Center, Bloomington, Indiana, United States